CLINICAL TRIAL: NCT01128634
Title: A Single-Centre, Randomised, Open-label Study to Evaluate the Effects of Steady-State Verapamil, a Moderate P-Glycoprotein and CYP3A4 Inhibitor, on the Pharmacokinetics of GSK573719 and GSK573719 in Combination With GW642444
Brief Title: Pharmacokinetic and Safety of GSK573719 and GW642444 Administered Individually and Concurrently, With Verapamilin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 113950
Record Dates: First submitted 2010-05-20; First posted 2010-05-24 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Verapamil; Anticholinergic, β2 agonist; P-GP; LABA; Muscarinic Receptor Antagonist; LAMA
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — GSK573719

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK573719 (Other): GSK573719
  Interventions: Drug: GSK573719
- GSK573719/GW642444 (Other): GSK573719/GW642444
  Interventions: Drug: GW573719/GW573719

INTERVENTIONS:
Drug: GSK573719 — 13 days dosing with GSK573719, once daily dosing from day 1 to 13, concurrent dosing with verapamil from day 9 to 13.
  Arms: GSK573719
Drug: GW573719/GW573719 — 13 days dosing with GSK573719/GW573719, once daily dosing from day 1 to 13, concurrent dosing with verapamil from day 9 to 13.
  Arms: GSK573719/GW642444

SUMMARY:
The purpose of this study is to see if the Pharmacokinetics and the Safety Profile of GSK573719 and GSK573719/GW642444 are effected by concurrent dosing with the PGP inhibitor verapamil.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin < 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: non childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy, double oophorectomy or bilateral salpingectomy., or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL and estradiol < 40 pg/ml (<140 pmol/L) or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until completion of the follow up visit.
* Body weight > 45 kg and BMI within the range 18 - 28 kg/m2 (inclusive).
* Capable of giving written informed consent and a signed and dated written informed consent is obtained, which includes compliance with the requirements and restrictions listed in the consent form.
* Normal spirometry (FEV1 ≥ 80% of predicted, FEV1/FVC ≥ 70%).
* Non-smokers (never smoked or not smoking for >6 months with <10 pack years history (Pack years = (cigarettes per day smoked/20) x number of years smoked))
* Available to complete the study

Exclusion Criteria:

* Any clinically important abnormality identified at the screening medical assessment (physical examination/medical history), clinical laboratory tests, ECG (12-lead) or from 24hr Holter monitoring. If the Investigator and the GSK Medical Monitor agree that a finding is unlikely to introduce additional risk factors and will not interfere with the study procedures a subject can be included.
* A mean QTc(B) value at screening >450msec, or an ECG that is not suitable for QT measurements (e.g. LBBB or poorly defined termination of the T wave).
* A history of elevated resting blood pressure or a mean blood pressure higher than 140/90 mmHg at screening.
* A mean heart rate outside the range 40-90 bpm at screening.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates and benzodiazepines. The detection of drugs with a legitimate medical use would not necessarily be an exclusion to study participation. The detection of alcohol would not be an exclusion at screening but would need to be negative pre-dose and during the study.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome).
* A positive test for HIV antibody (if testing required by local SOP's).
* History of regular alcohol consumption within 3months of the study defined as:

an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.

* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, verapamil or components thereof, known allergy or hypersensitivity to milk protein or the excipients lactose monohydrate and MgSt, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* The subject is unable to use the novel dry powder inhaler correctly.
* The subject has a known allergy or hypersensitivity to ipratropium bromide, tiotropium, atropine and any of its derivatives.
* Any adverse reaction including immediate or delayed hypersensitivity to any β2 agonist or sympathomimetic drug,.
* Subject is kept under regulatory of judicial order in an institution.
* Subject is mentally or legally incapacitated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-03-04 (Actual); Primary Completion 2010-04-26 (Actual); Study Completion 2010-04-26 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of plasma and urine | 15 days

SECONDARY OUTCOMES:
General safety and tolerability endpoints: adverse events, heart rate, systolic and diastolic blood pressure, 12- lead ECG (QTc(B), QTc(F)) and clinical laboratory safety tests. 24hr Holter monitoring | From first dose on day 1 through to Follow Up visit

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Mehta R, Kelleher D, Preece A, Hughes S, Crater G. Effect of verapamil on systemic exposure and safety of umeclidinium and vilanterol: a randomized and open-label study. Int J Chron Obstruct Pulmon Dis. 2013;8:159-67. doi: 10.2147/COPD.S40859. Epub 2013 Mar 27. PMID 23569370
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 113950 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113950?search=study&search_terms=113950#rs
- Available data/document: Clinical Study Report: 113950 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113950 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113950 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113950 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113950 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113950 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113950 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register